CLINICAL TRIAL: NCT03001726
Title: Gastrectomy Plus Chemotherapy Versus Chemotherapy Alone for Advanced Gastric Cancer With a Single Non-curable Factor
Brief Title: To Observe the Efficacy and Safety by Comparing Chemotherapy(Docetaxel, Oxaliplatin Plus S1 ) Followed With Radical Resection Versus Chemotherapy Alone in Advanced Gastric Cancer With Single Non-curable Factor.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Tianshu Liu, Chairman for the department of oncology, Shanghai Zhongshan Hospital
Other Study IDs: NEO-REGATTA
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2016-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastrectomy; Oxaliplatin; S 1 (combination); Tegafur; Docetaxel

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Gastrectomy plus chemotherapy: In patients assigned to surgery followed by chemo- therapy, a total, distal, or proximal gastrectomy with metastasis dissection was done depending on tumour location.
  Interventions: Procedure: Gastrectomy; Drug: oxaliplatin; Drug: S1; Drug: Docetaxel
- chemotherapy alone: Patients received chemotherapy alone.All patients received oral S1 80 mg/m2 per day (80-120 mg/day total dose depending on the patient's body surface area as follows: <1.25 m2, 80 mg; 1.25-1.5 m2, 100 mg; and >1.5 m2, 120 mg) on days 1-21 of every 3-week cycle, oxaliplatin 100 mg/m2 on day 1 of every 3-week cycle and docetaxel 40mg/m2 on day 1 of every 3-weeks cycle.
  Interventions: Drug: oxaliplatin; Drug: S1; Drug: Docetaxel

INTERVENTIONS:
Procedure: Gastrectomy — In patients assigned to surgery followed by chemo- therapy, a total, distal, or proximal gastrectomy with metastasis dissection was done depending on tumour location.
  Groups: Gastrectomy plus chemotherapy
Drug: oxaliplatin — oxaliplatin 100 mg/m2
  Other Names: Eloxatin
Drug: S1 — S1 40mg/m2
  Other Names: tegafur
Drug: Docetaxel — docetaxel 40 mg/m2
  Other Names: Taxotere

SUMMARY:
Investigators assessed the effectiveness of conversional gastrectomy compared with chemotherapy alone following docetaxel, oxalipaltin and S1 therapy for advanced gastric cancer with a single non-curable factor.

DETAILED DESCRIPTION:
Palliative chemotherapy is still the standard of care for incurable advanced gastric cancer. Several retrospective, single institutional studies have shown that the addition of gastrectomy to chemotherapy might improve patient survival among patients with metastatic gastric cancer with a single non-curable factor. However, REGATTA trial, a phase 3, randomized controlled trial, concluded an opposite conclusion that gastrectomy followed by chemotherapy did not show any survival benefit compared with chemotherapy alone in advanced gastric cancer with a single non-curable factor. Interestingly, five patients initially assigned to chemotherapy alone in the study had got survival benefit form gastrectomy with curative intent because of complete disappear of all non-curable factors during chemotherapy. This finding raised the question as to conversional radical surgery following upfront chemotherapy could be a possible treatment option. We assessed the effectiveness of conversional radical surgery following docetaxel, oxalipaltin and S1 therapy for advanced gastric cancer with a single non-curable factor.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gastric cancer with a single non-curable factor
* A single non-curable factor was defined as hepatic metastasis (H1; two to four lesions of maximum diameter ≤5 cm and minimum diameter ≥1 cm); peritoneal metastasis (P1) in the diaphragm or peritoneum caudal to the transverse colon without massive ascites or intestinal obstruction; positive cytology (CY1) when the cancer cells were found in the peritoneal washing; para-aortic lymph node (PAN) metastasis above the coeliac axis or below the inferior mesenteric artery (lymph node 16a1/b2 of maximum diameter ≥1 cm), or both; or ovary implant metastasis for one site or two.

Exclusion Criteria:

* Patients who can have radical resection.
* Patietns who have more than one metastasis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical diagnosis of gastric cancer with a single non-curable factor
Sampling Method: Non-Probability Sample
Enrollment: 228 (Estimated)
Dates: Start 2017-01; Primary Completion 2022-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | through study completion, an average of 2 year

SECONDARY OUTCOMES:
progression-free survival | through study completion, an average of 1 year

OTHER OUTCOMES:
response rate | through study completion, an average of 24 weeks
adverse events | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tianshu Liu, Physician, Principal Investigator — Zhongshan Hopital
Locations (1):
- Zhongshan hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cui Y, Yu Y, Zheng S, Ying J, Du Y, Wang Y, Wang X, Shen Z, Liu F, Lv M, Sun Y, Liu T. Does resection after neoadjuvant chemotherapy of docetaxel, oxaliplatin, and S-1 (DOS regimen) benefit for gastric cancer patients with single non-curable factor? a multicenter, prospective cohort study (Neo-REGATTA). BMC Cancer. 2023 Apr 4;23(1):308. doi: 10.1186/s12885-023-10773-x. PMID 37016303